CLINICAL TRIAL: NCT05149781
Title: Standardized Diagnosis and Treatment of Endocrine Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Endocrine Hypertension
MeSH Terms: interventions — Therapeutics; Antihypertensive Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, adrenal adenoma tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with EH: patients with endocrine hypertension
  Interventions: Procedure: Standardized diagnosis and treatment
- patients with PH: patients with primary hypertension

INTERVENTIONS:
Procedure: Standardized diagnosis and treatment — Patients with endocrine hypertension undergo surgery or medication depending on the cause after completion of standard diagnostic procedures. Patients with primary hypertension receive medication.
  Other Names: antihypertensive drugs
  Groups: patients with EH

SUMMARY:
Cases of endocrine hypertension or primary hypertension who have signed informed consent will be collected. Patients with endocrine hypertension will be divided into surgical treatment group and drug treatment group according to actual treatment situation. A database will be established for all patients. The investigators will comprehensively evaluate the general conditions, past medical history, metabolic and biochemical indicators, psychological status, cardiovascular risk factors. All the patients will be followed up for 12 months at baseline, 6 months and 12 months. Clinical data and specimen will be collected.

DETAILED DESCRIPTION:
The investigators will collect 100 patients with secretory hypertension and 100 patients with essential hypertension. Patients with endocrine hypertension will be divided into surgical treatment group and drug treatment group according to actual treatment situation. Resected specimens from surgical patients will be used for immunohistochemistry and western blot. A database will be established for all patients to assess their general situation, past medical history, metabolic and biochemical indicators, psychological status, cardiovascular risk factors, etc. The investigators expect to find more accurate screening indicators from blood and urine specimens. All the patients will be followed up for 12 months at baseline, 6 months and 12 months. Blood pressure, degree of atherosclerosis, biochemical markers, hormone levels and cardiac function indicators will be measured at three time points.

ELIGIBILITY:
Inclusion Criteria:

age≥18 years

Exclusion Criteria:

1. myocardial infarction
2. congestive heart failure
3. stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endocrine hypertension or primary hypertension treated at Affiliated Hospital of Nantong University between 2021 and 2024
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The control rate of blood pressure | 12 months
  The investigators will compare the proportion of patients with blood pressure below 140/90 mmHg after different treatments.

SECONDARY OUTCOMES:
Changes of carotid imima-media thickness | 12 months
  Carotid ultrasound will be used to observe the changes of carotid intima-media thickness after different treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gu Yunjuan, M.D/Ph.D, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Gu Yunjuan, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided